CLINICAL TRIAL: NCT03673332
Title: Elderly Cancer PatIents Treated for Advanced or Metastatic Melanoma or NSCLC, Safety and qualiTy of Life Under immunOtheraPies: a Phase IV Trial
Brief Title: Elderly Cancer PatIents, Safety and qualiTy of Life Under immunOtheraPies
Acronym: EPITOP-01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Société Francophone d'Onco-Gériatrie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPITOP-01-IPC 2017-049; 2018-002092-18 (EudraCT Number)
Record Dates: First submitted 2018-08-21; First posted 2018-09-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced or Metastatic Melanoma; Advanced or Metastatic NSCLC
Keywords: Elderly cancer patients; Immunotherapies
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This is a national prospective phase 4, multi-centre, single arm, open-label cohort study to evaluate the safety and efficacy of immune checkpoint inhibitors-based therapies in elderly patients with advanced or metastatic melanoma or NSCLC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment including immune checkpoint inhibitors (Experimental): All patients included in this study will receive approved immune-checkpoint inhibitors therapies, such as CTLA-4, PD-1, and PD-L1 inhibitors.
  Interventions: Drug: immune-checkpoint inhibitors therapies

INTERVENTIONS:
Drug: immune-checkpoint inhibitors therapies — All patients included in this study will receive approved immune-checkpoint inhibitors therapies, such as CTLA-4, PD-1, and PD-L1 inhibitors.

SUMMARY:
The co-primary objectives will be to assess the safety and quality of life under treatment.

DETAILED DESCRIPTION:
The co-primary objectives will be to assess the safety and quality of life under treatment. Secondary objectives will be evaluations of geriatric data modifications under treatment, efficacy (progression-free survival and overall survival), correlation between toxicity and efficacy, and comparison of the safety profiles between various immunotherapy regimens.

Another secondary objective will be the comparison between patients and clinicians symptom reporting. The investigators will also perform a pharmacokinetics analysis on PD1-monoclonal antibodies to improve the understanding of PD-1 inhibitors pharmacokinetics for the elderly population.

Finally, toxicity and efficacy will be compared to immunological parameters such as the description of tumor infiltrating lymphocytes, markers of immunosenescence and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to start a treatment including immune checkpoint inhibitors (Nivolumab, Ipilimumab, Pembrolizumab, and so on…)
* Diagnosis of advanced or metastatic melanoma or NSCLC (All treatment lines will be allowed)
* Age ≥ 70 years
* Having personally signed and dated informed consent
* Patient affiliated to the ''National security'' regimen or beneficiary of this regimen

Exclusion Criteria:

* Immune checkpoint inhibitor therapy initiated before study enrolment
* Concomitant participation in other investigational clinical trials involving an immune checkpoint inhibitor
* Immune checkpoint inhibitor treatment in a context of other solid tumours
* Immune checkpoint inhibitor treatment in a context of haematological malignancies
* Being unable or unwilling to comply with the requirements of the protocol, as assessed by the investigator
* Patient in urgency situation, adult under legal protection, or unable to give his consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Number of participants adverse events as assessed by CTCAE v5.0 | From treatment initiation to 18 weeks after treatment initiation. (up to 24 months)
  Description of adverse events' type, incidence, severity (CTCAE v.5.0), timing, seriousness, and relatedness. This endpoint will be based on the rate of grade ≥ 3 adverse events 18 weeks after treatment initiation, defined as medical assessment of safety including adverse events' type, incidence, severity (graded by the CTCAE] v. 5.0), timing, seriousness, and relatedness. This will include clinical as well as biological toxicities such as liver and endocrine dysfunctions. All high grade adverse events will be taken into account.
European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (QLQ-C30) and Elderly Cancer Patients module (QLQ - ELD14), combined to compute a total score (between 44 and 128 points) | From inclusion until 24 weeks after treatment initiation (up to 24 months)
  Quality of life will be evaluated using the EORTC QLQ-C30 and QLQ-ELD14 questionnaires collected at inclusion and at every treatment cycles during the first 6 weeks, then every 6 weeks until treatment discontinuation. The proportion of patients with a decrease superior or equal to 10% for their global score between baseline and at 24 weeks after treatment initiation will be estimated.

SECONDARY OUTCOMES:
geriatric data modifications under treatment | From inclusion until treatment discontinuation (up to 24 months)
  Geriatric data assessment will be done at inclusion and every 6 weeks until treatment discontinuation. Exhaustive data will be collected at inclusion. The investigators will also assess the G-CODE (Geriatric Core Dataset), a recently described minimum geriatric data set (see SOFOG guidelines). G-CODE assessment will be repeated every 6 weeks during treatment and at treatment discontinuation. These data will be collected either by the geriatrician or trained clinical research nurses during geriatric consultation as part of geriatric follow-up, an integral part of the patient management.
compare patients and clinician symptoms reporting | From treatment initiation to 18 weeks after treatment initiation.(up to 24 months)
  Reminder of CTCAE version 5.0 will be completed by clinicians before every treatment cycle. Patients will also complete a language adapted version of patient-reported outcome PRO-CTCAE questionnaire. For all symptoms, the investigators will measure the proportion of pairs for which clinicians and patients gave an identical grade. The investigators will also measure the proportion of pairs that will disagree for each symptom by one point (e.g., patient grade 2 and clinician grade 1), and the proportion that will disagree by two or more points (e.g., patient grade 2 and clinician grade 4). The investigators will also record the number of symptoms for which each pair agreed.
Progression-free survival | time from treatment beginning to radiological or clinical progression of the disease, or death of any cause. (up to 24 months)
  Evaluation of Progression-free Survival (PFS) will be defined as the time from treatment beginning to radiological (according to the RECIST 1.1 criteria) or clinical progression of the disease as declared by the investigators, or death of any cause. Radiological evaluations will be performed every 6 weeks.
Overall Survival | time from treatment beginning to death of any cause (up to 24 months)
  Overall Survival (OS) will be defined as the time from treatment beginning to death of any cause.
correlation between toxicity and efficacy | time from treatment beginning to radiological or clinical progression of the disease, or death of any cause. (up to 24 months)
  Correlation between occurrence of auto-immune adverse events (with a landmark time at week 18) and efficacy (PFS).
rate of grade 3 to 5 adverse events 18 weeks after treatment initiation | From treatment initiation to 18 weeks after treatment initiation.(up to 24 months)
  Safety profiles comparison according to treatment regimen (PD1-inhibitor monotherapy vs PD1- inhibitor/CTLA4-inhibitor combination vs CTLA-inhibitor monotherapy vs PDL1-inhibitor if available at time of trial beginning) will be performed by looking at the rate of grade 3 to 5 adverse events 18 weeks after treatment initiation for each therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Sabatier, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (9):
- France (9):
  - Assistance Publique des Hôpitaux de Marseille, Marseille, Bouches Du Rhône
  - Institut Paoli-Calmettes, Marseille, Bouches-du Rhône
  - Institut BERGONIE, Bordeaux
  - CENTRE Francois Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Institut Du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut De Cancérologie de l'Ouest, Saint-Herblain
  - IUCT-Oncopole Institut Claudius Rigaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balducci L, Extermann M. Management of cancer in the older person: a practical approach. Oncologist. 2000;5(3):224-37. doi: 10.1634/theoncologist.5-3-224. PMID 10884501
- [Background] Basch E, Iasonos A, McDonough T, Barz A, Culkin A, Kris MG, Scher HI, Schrag D. Patient versus clinician symptom reporting using the National Cancer Institute Common Terminology Criteria for Adverse Events: results of a questionnaire-based study. Lancet Oncol. 2006 Nov;7(11):903-9. doi: 10.1016/S1470-2045(06)70910-X. PMID 17081915
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Cella D, Grunwald V, Nathan P, Doan J, Dastani H, Taylor F, Bennett B, DeRosa M, Berry S, Broglio K, Berghorn E, Motzer RJ. Quality of life in patients with advanced renal cell carcinoma given nivolumab versus everolimus in CheckMate 025: a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):994-1003. doi: 10.1016/S1470-2045(16)30125-5. Epub 2016 Jun 6. PMID 27283863
- [Background] Champiat S, Dercle L, Ammari S, Massard C, Hollebecque A, Postel-Vinay S, Chaput N, Eggermont A, Marabelle A, Soria JC, Ferte C. Hyperprogressive Disease Is a New Pattern of Progression in Cancer Patients Treated by Anti-PD-1/PD-L1. Clin Cancer Res. 2017 Apr 15;23(8):1920-1928. doi: 10.1158/1078-0432.CCR-16-1741. Epub 2016 Nov 8. PMID 27827313
- [Background] Daste A, Domblides C, Gross-Goupil M, Chakiba C, Quivy A, Cochin V, de Mones E, Larmonier N, Soubeyran P, Ravaud A. Immune checkpoint inhibitors and elderly people: A review. Eur J Cancer. 2017 Sep;82:155-166. doi: 10.1016/j.ejca.2017.05.044. Epub 2017 Jul 6. PMID 28689093
- [Background] Du-Thanh A, Lesage C, Ferreira E, Dereure O, Guillot B. [Innovative therapies for metastatic melanoma in elderly patients]. Ann Dermatol Venereol. 2015 Oct;142(10):549-56. doi: 10.1016/j.annder.2015.03.022. Epub 2015 May 16. French. PMID 25986740
- [Background] Extermann M. Measurement and impact of comorbidity in older cancer patients. Crit Rev Oncol Hematol. 2000 Sep;35(3):181-200. doi: 10.1016/s1040-8428(00)00090-1. PMID 10960800
- [Background] Fitzsimmons D, Gilbert J, Howse F, Young T, Arrarras JI, Bredart A, Hawker S, George S, Aapro M, Johnson CD. A systematic review of the use and validation of health-related quality of life instruments in older cancer patients. Eur J Cancer. 2009 Jan;45(1):19-32. doi: 10.1016/j.ejca.2008.07.036. Epub 2008 Sep 25. PMID 18823775
- [Background] Greenhalgh J. The applications of PROs in clinical practice: what are they, do they work, and why? Qual Life Res. 2009 Feb;18(1):115-23. doi: 10.1007/s11136-008-9430-6. Epub 2008 Dec 23. PMID 19105048
- [Background] Helissey C, Vicier C, Champiat S. The development of immunotherapy in older adults: New treatments, new toxicities? J Geriatr Oncol. 2016 Sep;7(5):325-33. doi: 10.1016/j.jgo.2016.05.007. Epub 2016 Jun 16. PMID 27318796
- [Background] Hjermstad MJ, Fayers PM, Bjordal K, Kaasa S. Using reference data on quality of life--the importance of adjusting for age and gender, exemplified by the EORTC QLQ-C30 (+3). Eur J Cancer. 1998 Aug;34(9):1381-9. doi: 10.1016/s0959-8049(98)00136-1. PMID 9849421
- [Background] Hua C, Boussemart L, Mateus C, Routier E, Boutros C, Cazenave H, Viollet R, Thomas M, Roy S, Benannoune N, Tomasic G, Soria JC, Champiat S, Texier M, Lanoy E, Robert C. Association of Vitiligo With Tumor Response in Patients With Metastatic Melanoma Treated With Pembrolizumab. JAMA Dermatol. 2016 Jan;152(1):45-51. doi: 10.1001/jamadermatol.2015.2707. PMID 26501224
- [Background] Ishida Y, Agata Y, Shibahara K, Honjo T. Induced expression of PD-1, a novel member of the immunoglobulin gene superfamily, upon programmed cell death. EMBO J. 1992 Nov;11(11):3887-95. doi: 10.1002/j.1460-2075.1992.tb05481.x. PMID 1396582
- [Background] Khoja L, Day D, Wei-Wu Chen T, Siu LL, Hansen AR. Tumour- and class-specific patterns of immune-related adverse events of immune checkpoint inhibitors: a systematic review. Ann Oncol. 2017 Oct 1;28(10):2377-2385. doi: 10.1093/annonc/mdx286. PMID 28945858
- [Background] Lafage-Pochitaloff M, Costello R, Couez D, Simonetti J, Mannoni P, Mawas C, Olive D. Human CD28 and CTLA-4 Ig superfamily genes are located on chromosome 2 at bands q33-q34. Immunogenetics. 1990;31(3):198-201. doi: 10.1007/BF00211556. PMID 2156778
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Manoussakis MN, Tzioufas AG, Silis MP, Pange PJ, Goudevenos J, Moutsopoulos HM. High prevalence of anti-cardiolipin and other autoantibodies in a healthy elderly population. Clin Exp Immunol. 1987 Sep;69(3):557-65. PMID 3499270
- [Background] Michelson H, Bolund C, Brandberg Y. Multiple chronic health problems are negatively associated with health related quality of life (HRQoL) irrespective of age. Qual Life Res. 2000;9(10):1093-104. doi: 10.1023/a:1016654621784. PMID 11401042
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Background] Naidoo J, Page DB, Li BT, Connell LC, Schindler K, Lacouture ME, Postow MA, Wolchok JD. Toxicities of the anti-PD-1 and anti-PD-L1 immune checkpoint antibodies. Ann Oncol. 2015 Dec;26(12):2375-91. doi: 10.1093/annonc/mdv383. Epub 2015 Sep 14. PMID 26371282
- [Background] Nghiem PT, Bhatia S, Lipson EJ, Kudchadkar RR, Miller NJ, Annamalai L, Berry S, Chartash EK, Daud A, Fling SP, Friedlander PA, Kluger HM, Kohrt HE, Lundgren L, Margolin K, Mitchell A, Olencki T, Pardoll DM, Reddy SA, Shantha EM, Sharfman WH, Sharon E, Shemanski LR, Shinohara MM, Sunshine JC, Taube JM, Thompson JA, Townson SM, Yearley JH, Topalian SL, Cheever MA. PD-1 Blockade with Pembrolizumab in Advanced Merkel-Cell Carcinoma. N Engl J Med. 2016 Jun 30;374(26):2542-52. doi: 10.1056/NEJMoa1603702. Epub 2016 Apr 19. PMID 27093365
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Robert C, Karaszewska B, Schachter J, Rutkowski P, Mackiewicz A, Stroiakovski D, Lichinitser M, Dummer R, Grange F, Mortier L, Chiarion-Sileni V, Drucis K, Krajsova I, Hauschild A, Lorigan P, Wolter P, Long GV, Flaherty K, Nathan P, Ribas A, Martin AM, Sun P, Crist W, Legos J, Rubin SD, Little SM, Schadendorf D. Improved overall survival in melanoma with combined dabrafenib and trametinib. N Engl J Med. 2015 Jan 1;372(1):30-9. doi: 10.1056/NEJMoa1412690. Epub 2014 Nov 16. PMID 25399551
- [Background] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, Lebbe C, Baurain JF, Testori A, Grob JJ, Davidson N, Richards J, Maio M, Hauschild A, Miller WH Jr, Gascon P, Lotem M, Harmankaya K, Ibrahim R, Francis S, Chen TT, Humphrey R, Hoos A, Wolchok JD. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med. 2011 Jun 30;364(26):2517-26. doi: 10.1056/NEJMoa1104621. Epub 2011 Jun 5. PMID 21639810
- [Background] Solana R, Tarazona R, Gayoso I, Lesur O, Dupuis G, Fulop T. Innate immunosenescence: effect of aging on cells and receptors of the innate immune system in humans. Semin Immunol. 2012 Oct;24(5):331-41. doi: 10.1016/j.smim.2012.04.008. Epub 2012 May 4. PMID 22560929
- [Background] Wheelwright S, Darlington AS, Fitzsimmons D, Fayers P, Arraras JI, Bonnetain F, Brain E, Bredart A, Chie WC, Giesinger J, Hammerlid E, O'Connor SJ, Oerlemans S, Pallis A, Reed M, Singhal N, Vassiliou V, Young T, Johnson C. International validation of the EORTC QLQ-ELD14 questionnaire for assessment of health-related quality of life elderly patients with cancer. Br J Cancer. 2013 Aug 20;109(4):852-8. doi: 10.1038/bjc.2013.407. Epub 2013 Jul 18. PMID 23868003
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Bandeen-Roche K, Xue QL, Ferrucci L, Walston J, Guralnik JM, Chaves P, Zeger SL, Fried LP. Phenotype of frailty: characterization in the women's health and aging studies. J Gerontol A Biol Sci Med Sci. 2006 Mar;61(3):262-6. doi: 10.1093/gerona/61.3.262. PMID 16567375
- [Background] Davis HS, MacPherson K, Merry HR, Wentzel C, Rockwood K. Reliability and validity of questions about exercise in the Canadian Study of Health and Aging. Int Psychogeriatr. 2001;13 Supp 1:177-82. doi: 10.1017/s1041610202008128. PMID 11892965
- [Background] Cornali C, Franzoni S, Frisoni GB, Trabucchi M. Anorexia as an independent predictor of mortality. J Am Geriatr Soc. 2005 Feb;53(2):354-5. doi: 10.1111/j.1532-5415.2005.53126_4.x. No abstract available. PMID 15673368
- [Background] Cheng ST, Chan AC. Comparative performance of long and short forms of the Geriatric Depression Scale in mildly demented Chinese. Int J Geriatr Psychiatry. 2005 Dec;20(12):1131-7. doi: 10.1002/gps.1405. PMID 16315157
- [Background] Clement JP, Nassif RF, Leger JM, Marchan F. [Development and contribution to the validation of a brief French version of the Yesavage Geriatric Depression Scale]. Encephale. 1997 Mar-Apr;23(2):91-9. French. PMID 9264935
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Borson S, Scanlan JM, Chen P, Ganguli M. The Mini-Cog as a screen for dementia: validation in a population-based sample. J Am Geriatr Soc. 2003 Oct;51(10):1451-4. doi: 10.1046/j.1532-5415.2003.51465.x. PMID 14511167
- [Background] Borson S, Scanlan J, Brush M, Vitaliano P, Dokmak A. The mini-cog: a cognitive 'vital signs' measure for dementia screening in multi-lingual elderly. Int J Geriatr Psychiatry. 2000 Nov;15(11):1021-7. doi: 10.1002/1099-1166(200011)15:113.0.co;2-6. PMID 11113982
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Barberger-Gateau P, Dartigues JF, Letenneur L. Four Instrumental Activities of Daily Living Score as a predictor of one-year incident dementia. Age Ageing. 1993 Nov;22(6):457-63. doi: 10.1093/ageing/22.6.457. PMID 8310892
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222